CLINICAL TRIAL: NCT05690308
Title: A Novel Training Method to Reduce Fall Risk in People with Parkinson's Disease: the Role of the Balance Organ
Brief Title: Visual Perturbation Training to Reduce Fall Risk in People with Parkinson's Disease
Acronym: Vesti-PD
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Ghent (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: ONZ-2022-0404
Record Dates: First submitted 2022-09-01; First posted 2023-01-19 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-09

CONDITIONS: Parkinson Disease; Vestibular Disorder; Gait; Falling
Keywords: Virtual reality
MeSH Terms: conditions — Parkinson Disease; Vestibular Diseases

STUDY DESIGN:
Intervention Model Description: Randomized Controlled Trial
Who Masked: Participant
Masking Description: Participants will not be informed if they are allocated to the experimental intervention or the control 'sham' intervention.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Experimental visual perturbation treadmill training (Experimental): Participants assigned to the experimental intervention will receive 6 weeks, 2x per week of visual perturbation treadmill training using the GRAIL system. This will consist of maximum 30 minutes of walking on the treadmill while translations and rotations of the projected environment are applied.
  Interventions: Other: Visual perturbation treadmill training
- Control treadmill training (Sham Comparator): Participants assigned to the control intervention will receive 6 weeks, 2x per week of treadmill only training. This will consist of maximum 30 minutes of walking on the treadmill without any visual perturbations.
  Interventions: Other: Regular treadmill training

INTERVENTIONS:
Other: Visual perturbation treadmill training — 12 sessions of (max 30 minutes) walking at comfortable speed on an instrumented treadmill in a virtual reality environment (Gait Real-time Analysis Interactive Lab system, MOTEK) with projected visual perturbations.
  Arms: Experimental visual perturbation treadmill training
Other: Regular treadmill training — 12 sessions of (max 30 minutes) walking at comfortable speed on an instrumented treadmill
  Arms: Control treadmill training

SUMMARY:
Falls during walking are common in people with Parkinson's Disease (PD). Fall risk can be attributed in part to the loss of automaticity in walking and an increased reliance on sensory cues, such as the input from the balance organ. In this project the investigators want to assess the effectiveness of rehabilitation training aiming to improve this vestibular input. The effects of a visual perturbation training in a virtual reality environment will be compared to conventional treadmill training.

DETAILED DESCRIPTION:
Fifty participants (50-65 years) with idiopathic PD (Hoehn & Yahr scale 2-3) will be randomly assigned to the intervention group receiving four weeks of VPT in a VR environment using the Gait Real-time Analysis Interactive Lab system (GRAIL) or a control group receiving four weeks of regular treadmill training. Primary outcome measures are spatio-temporal outcome parameters of gait and dynamic stability (gait speed, stride time/length, cadence, step-to-step variability, step width variability and trunk sway), and self-reported falls, and will be recorded at all testing phases (pre-test, after baseline, after intervention and after detraining). Secondary outcome measures will include assessments of central and peripheral vestibular function (Cervical and ocular Vestibular Evoked Myogenic Potentials) for correlation with the primary outcome measures. The secondary outcomes will be recorded at pre-testing and directly after the intervention phase.

ELIGIBILITY:
Inclusion Criteria:

* Idiopathic Parkinson's disease
* Aged between 50-65 years
* Bilateral symptoms
* Able to walk unassisted for 20 minutes (Hoehn & Yahr stage II-III)
* Stable medication dosage (if any)
* No cognitive disablity

Exclusion Criteria:

* Non-idiopathic Parkinson's disease
* Strong variation in expressed symptoms
* Inability to walk unassisted for 20 minutes
* Underwent a medical procedure to treat Parkinson symptoms (e.g. duodopa pump, deep brain stimulator)
* Cognitive disability (score < 21 on the Montreal Cognitive Assessment)
* Illness other than Parkinson's disease (flu, Covid-19) or disabilities that may affect gait or equilibrium
* Clogged ear(s)
* Regular fainting episodes
* Weight over 120 kg
* Participation in other clinical studies

Ages: 50 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 35 (Actual)
Dates: Start 2022-12-20 (Actual); Primary Completion 2024-03-30 (Actual); Study Completion 2024-05-13 (Actual)

PRIMARY OUTCOMES:
Change from baseline in gait speed after 6 weeks training | Week 1 to week 6 of training intervention
  Delta in average gait speed in m/s
Change from baseline in cadence after 6 weeks training | Week 1 to week 6 of training intervention
  Delta in steps per minute
Change from baseline in stride time after 6 weeks training | Week 1 to week 6 of training intervention
  Delta in average duration (+variability) of a single step in ms
Change from baseline in step length after 6 weeks training | Week 1 to week 6 of training intervention
  Delta in average length (+variability) of a single step in cm
Change from baseline in step width after 6 weeks training | Week 1 to week 6 of training intervention
  Delta in average width(+variability) of a single step in cm
Change from baseline in trunk sway after 6 weeks training | Week 1 to week 6 of training intervention
  Delta in medio-lateral and anterior-posterior movement of the center of mass as determined using 3D motion capturing in cm

SECONDARY OUTCOMES:
Assessments of central and peripheral vestibular function | Pre-test 1 at start of the study
  Cervical and ocular vestibular evoked myogenic potentials
Assessments of central and peripheral vestibular function | Post-test within 1 week after conclusion of the training intervention
  Cervical and ocular vestibular evoked myogenic potentials
Self-reported falls | Monthly up to six months after last training
  Falls recorded in fall diary

OTHER OUTCOMES:
Assessment of fear of falling | Pre-test 2 at start of the study
  Fear of falling recorded using the Iconographical Falls Efficacy Scale
Assessment of fear of falling | Post-test within 1 week after conclusion of the training intervention
  Fear of falling recorded using the Iconographical Falls Efficacy Scale

CONTACTS AND LOCATIONS:
Overall Officials: Patrick Santens, Prof., Principal Investigator — UZ Gent
Locations (1):
- UZ Gent, Ghent, East-Flanders, Belgium

IPD SHARING:
Plan to Share IPD: No